CLINICAL TRIAL: NCT06832254
Title: Effectiveness of Cryotherapy Versus Dexamethasone on Reducing Postoperative Pain in Permanent Mandibular Molars with Irreversible Pulpitis: a Randomized Controlled Clinical Trial
Brief Title: Cryotherapy Versus Dexamethasone on Postoperative Pain in Permanent Mandibular Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13.02.2025/151
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Pulpitis - Irreversible
Keywords: Cryotherapy; Irrevesible pulpitis; Dexamethasone; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cryotherapy; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Irrigation was performed with a 30 G navitip needle and 2.5% sodium hypochlorite (NaOCl). A total of 11 mL of NaOCl was used in each root canal, 2 mL after coronal preparation, 2 mL after middle third preparation, 2 mL after apical third preparation and 5 mL in the final irrigation. After irrigation with NaOCl, each root canal was irrigated with 2 mL saline, 2 mL 17% EDTA and finally all canals were irrigated with a total of 20 mL of normal saline for 5 minutes.
- Cryotherapy Group (Experimental): Irrigation was performed with a 30 G navitip needle and 2.5% sodium hypochlorite (NaOCl). A total of 11 mL of NaOCl was used in each root canal, 2 mL after coronal preparation, 2 mL after middle third preparation, 2 mL after apical third preparation and 5 mL in the final irrigation. After irrigation with NaOCl, each root canal was irrigated with 2 mL saline, 2 mL 17% EDTA and finally all canals were irrigated with a total of 20 mL of cold (2 °C) saline for 5 minutes.
  Interventions: Other: Cryotherapy
- Dexamethasone Group (Experimental): Irrigation was performed with a 30 G navitip needle and 2.5% sodium hypochlorite (NaOCl). A total of 11 mL of NaOCl was used in each root canal, 2 mL after coronal preparation, 2 mL after middle third preparation, 2 mL after apical third preparation and 5 mL in the final irrigation. After irrigation with NaOCl, each root canal was irrigated with 2 mL saline, 2 mL 17% EDTA, 2 mL saline and 1 mL dexamethasone.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Other: Cryotherapy — The root canals were irrigated with 2 °C saline solution in final irrigation in cryotherapy group.
  Arms: Cryotherapy Group
Drug: Dexamethasone — Each root canal was irrigated with 1 mL dexamethasone solution in final irrigation in dexamethasone group.
  Arms: Dexamethasone Group

SUMMARY:
The goal of this clinical trial was to evaluate cryotherapy versus dexamethasone on the intensity of postoperative pain in root canal treatment procedures in mandibular first molar teeth with symptomatic irreversible pulpitis. The main question it aims to answer is:

* Does controlled irrigation with cold saline in root canal treatment reduce the severity of postoperative pain?
* Does controlled irrigation with dexamethasone in root canal treatment reduce the severity of postoperative pain? In the cryotherapy group, unlike the control and dexamethasone group, the root canals were irrigated with 2 °C salin solution in final irrigation.

In the dexamethasone group, unlike the control and cryotherapy group, the root canals were irrigated with 1 mL dexamethasone solution in final irrigation.

ELIGIBILITY:
Inclusion Criteria:

* Vital mandibular first and second molars with 3 root canals that responded positively to the cold test and electric pulp test
* Patients who had not taken analgesics or antibiotics in the last 24 hours before the procedure were included in the study.

Exclusion Criteria:

* Devital mandibular first and second molars that responded negatively to cold tests and electric pulp tests
* Mandibular first and second molars with poor periodontal status (pocket depth > 4 mm),
* Mandibular first and second molars with 4 or more root canals detected radiographically or after opening the endodontic access cavity were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to 72 hours
  The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain (10) imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Koray Yılmaz, DDS MSc, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers MJ, Johnson BR, Remeikis NA, BeGole EA. Comparison of effect of intracanal use of ketorolac tromethamine and dexamethasone with oral ibuprofen on post treatment endodontic pain. J Endod. 1999 May;25(5):381-4. doi: 10.1016/S0099-2399(06)81176-3. PMID 10530266
- [Background] Solomon RV, Paneeru SP, Swetha C, Yatham R. Comparative evaluation of effect of intracanal cryotherapy and corticosteroid solution on post endodontic pain in single visit root canal treatment. J Clin Exp Dent. 2024 Mar 1;16(3):e250-e256. doi: 10.4317/jced.61023. eCollection 2024 Mar. PMID 38600937
- [Background] Dildar I, Moghal A, Mirza A, Zaheer MA, Mallick MR, Munir S. Evaluation of Postoperative Pain after Using Dexamethasone Intracanal Rinse in Irreversible Pulpitis. J Coll Physicians Surg Pak. 2024 Apr;34(4):390-393. doi: 10.29271/jcpsp.2024.04.390. PMID 38576278